CLINICAL TRIAL: NCT05208593
Title: Alcohol Protective Behavioral Strategies and Thinking About the Past
Brief Title: Alcohol PBS and Thinking About the Past
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: University of Central Florida (Other)
Responsible Party: Principal Investigator, Sherecce A Fields, Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB20201070D
Record Dates: First submitted 2021-09-14; First posted 2022-01-26 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Drinking in College
MeSH Terms: conditions — Alcohol Drinking in College

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Negative Event Only (Placebo Comparator): Participants will be asked to think of a specific example of the most (or one of the most) negative, unpleasant event with alcohol they have experienced; the event they choose must have occurred at least a year ago. Or they will be asked to think of the most significant event that has occurred in the past year. After thinking of a specific event, they will be given three minutes to write about their experience. The writing prompt will ask that they express the event information in a few sentences. This writing prompt will help participants place themselves back into that moment and access salient emotions and cognition about it. Similar negative event prompts have been used in counterfactual thinking studies (McFarland & Alvaro, 2000; White & Lehman, 2005).
  Interventions: Behavioral: Negative Event Only
- Negative Event + Factual Thinking Task (Active Comparator): Participants in this group, the event plus the factual thinking task condition, will be told the following after completing the negative event writing task, "After disappointing and/or negative experiences like the one you described on the previous page, people often think about the details of the situation. For example, when it happened, who was involved, and what happened right before or after the incident occurred. In the space below please provide examples of some of these details.." There will be 10 blank boxes below the instructions and participants will be asked to provide some examples of details from their traumatic event. They will be asked to only list as many as they can naturally recall without repeating any. This procedure is derived from Kray and colleague's (2010) study on counterfactual thinking and meaning in life.
  Interventions: Behavioral: Negative Event + Factual Thinking Task
- Negative Event + Counterfactual Task (Experimental): Participants will be told after completing the negative event writing task, "After disappointing and/or negative experiences like the one you described, people sometimes cannot help thinking "what if…" or "if only…" and imagining how things might have gone differently. That is, if only I had done something differently, the negative drinking situation could have been avoided or turned out better. In the box below please identify things that, had they been different, would have improved the outcome of the negative drinking situation you described earlier and briefly describe how the outcome would have been better." Participants will be asked to list three counterfactuals about the event. Participants will also be asked to think of situations where these strategies could be used, to list out any obstacles that might prevent them from implementing these strategies and to indicate their intention to use each strategy over the next week.
  Interventions: Behavioral: Negative Event + Counterfactual Task
- Personalized Normative Feedback (Experimental): Participants in this group, the personalized normative feedback, will be asked to rate the frequency and quantity of TAMU students that use PBS when drinking.
  Interventions: Behavioral: Personalized Normative Feedback

INTERVENTIONS:
Behavioral: Negative Event + Counterfactual Task — Participants will complete a counterfactual based intervention where they come up with three if only..then statements about how a past drinking behavior could have been altered to be better and to think about protective behavioral strategies that they could use in a future similar situation to make the outcome better.
  Arms: Negative Event + Counterfactual Task
Behavioral: Personalized Normative Feedback — Participants will be asked to rate the frequency and quantity of students who use protective behavioral strategies while drinking. They will be given feedback on how close their estimate is from the national averages.
  Arms: Personalized Normative Feedback
Behavioral: Negative Event + Factual Thinking Task — Active Control condition where participants write about a negative event and list three facts about it
  Arms: Negative Event + Factual Thinking Task
Behavioral: Negative Event Only — Participants are asked to write about a negative event related to alcohol and write about it
  Arms: Negative Event Only

SUMMARY:
Individuals often think of how a situation or outcome could have turned out differently -- if only something was different or something had changed, then the outcome could have been better or worse. This is a common type of thinking, known as counterfactual thinking, that often takes the form of "if only" statements. These thoughts are frequent after negative events, but have also been found to occur after positive events and 'near misses'. Research has shown that their evaluative nature elicits a variety of consequences, such as biased decision making, changes in an event's meaningfulness, heightened positive or negative affect, and future behavioral changes (such as intentions, motivation, persistence/effort. Specifically, many areas of research involving counterfactuals have often looked into key elements that are often discussed in other health behavior literature, such as self-efficacy, motivation, and intentions. One such area that incorporates these elements is health promotion literature, such as Protective Behavioral Strategies (PBS) and alcohol consumption. The objectives of this study are laid out as such: First, to further explore the role counterfactuals play in increasing an individual's intentions toward behavioral change. Second, to further elucidate the inner and outer workings of Protective Behavioral Strategies for increasing positive health behaviors. Finally, to address the applicability of a counterfactual intervention on promoting intentions to use PBS.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years

Exclusion Criteria:

* no exclusions at baseline
* participants who do not follow the instructions for the specific writing task will be unable to sign-up for the remaining follow up sessions (Parts 2-6) and will be excluded the final data analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Protective Behavioral Strategies-20 | Weeks 1 - 6
  The Protective Behavioral Strategy-20 measure is a 20-item questionnaire assessing the use of three types of Protective Behavioral Strategies: serious harm reduction (8 items), stopping/limiting drinking (7 items), and manner of drinking (5 items). Each item has response options consisting of 1 (Never), 2 (Rarely), 3 (Occasionally), 4 (Sometimes), 5 (Usually), 6 (Always); there is also a Do not wish to respond option. Protective Behavioral Strategy Use scores are average scores for each subscale, with minimum scores of 0 and maximum scores of 6. Higher scores indicate greater use of protective behavioral strategies.
Young Adult Alcohol Consequences Questionnaire | Week 1
  The Young Adult Alcohol Consequences Questionnaire is a 48-item questionnaire assessing problems from alcohol consumption within the last three months. Each item is categorized into one of eight problem domains: social/interpersonal, academic/occupational, risky behavior, impaired control, poor self-care, diminished self-perception, blackout drinking, and physiological dependence. For each item, participants select Yes, No, or Do not wish to respond to indicate whether they have experienced each problem from alcohol consumption (e.g., "I have become very rude, obnoxious or insulting after drinking"). If a participant selects Yes that is indicative of the participant having experienced that specific consequence from alcohol consumption.
Alcohol Use Contemplation to Change Ladder | Week 1
  To assess an individual's contemplation to change their alcohol drinking behavior, a Contemplation to Change Ladder (Biener & Abrams, 1991) will be used. This ladder displays response options on a ladder graphic, with rungs starting at 0 and ending at 10; each rung increases by one point value as you go up the ladder. Anchors with text descriptions are located at points 0 (No thought of quitting), 2 (Think I need to consider quitting someday), 5 (Think I should quit but not quite ready), 8 (Starting to think about how to change my drinking patterns), and 10 (Taking action to quit e.g., cutting down, enrolling in a program). The higher a participant selects a rung on the ladder, the higher the contemplation to change their alcohol drinking behavior.
Change in Indication of Drinking and Strategy Use | Week 2 - Week 6
  A measure that assesses an individual's ability to avoid alcohol if they wanted to as well as binge-drinking or the ability to drink less in the next week

SECONDARY OUTCOMES:
Change in Perceived Behavioral Control | Week 1 and Week 2
  The Perceived Behavioral Control questionnaire measure is made up of six items. Three items assess the individual's ability to avoid alcohol if they wanted to and three items assess binge-drinking or the ability to drink less than 7(females) or 10 (males) units in a single session in the next week. Each item is scored on separate 7-point bipolar adjective scales (e.g., "For me to avoid drinking alcohol is…" very difficult to very easy). The six items will be averaged together to obtain an overall score for Perceived Behavioral Control. Higher scores indicate greater perceived behavioral control to control drinking behavior.
Change in Delay Discounting | Week 1, Week 4 and Week 6
  A measure of the amount participants discount delayed rewards
Change in Counterfactual Use and Intentions | Week 2 - Week 6
  Participants responses about whether they did counterfactuals in the past week and their intentions to use those behaviors in the next week.
Change in Personal Assessment of Responsible Drinker Identity Scale | Week 1, Week 4 and Week 6
  Participants are asked to indicate how true each statement in the Personal Assessment of Responsible Drinker Identity Scale is of the participant's experiences overall. Each item of this measure has response options ranging from 1 (not at all true) to 5 (completely true). Higher scores reflect greater agreement with identifying as a responsible drinker.
Change in Perceptions of Protective Behavioral Strategies | Week 1 - Week 6
  Questions about the percentage and frequency of use of protective behavioral strategies among college students.
Change in Contemplation to Change Ladder | Week 1 and Week 2
  To assess an individual's contemplation to change their alcohol drinking behavior, a Contemplation to Change Ladder (Biener & Abrams, 1991) will be used. This ladder displays response options on a ladder graphic, with rungs starting at 0 and ending at 10; each rung increases by one point value as you go up the ladder. Anchors with text descriptions are located at points 0 (No thought of quitting), 2 (Think I need to consider quitting someday), 5 (Think I should quit but not quite ready), 8 (Starting to think about how to change my drinking patterns), and 10 (Taking action to quit e.g., cutting down, enrolling in a program). The higher a participant selects a rung on the ladder, the higher the contemplation to change their alcohol drinking behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Dvorak, PhD, Principal Investigator — University of Central Florida; Rachel Smallman, PhD, Principal Investigator — Texas A&M University; Sherecce Fields, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ajzen, I., & Sheikh, S. (2013). Action versus inaction: Anticipated affect in the theory of planned behavior. Journal of Applied Social Psychology, 43(1), 155-162. https://doi.org/10.1111/j.1559-1816.2012.00989.x
- [Background] Cooke R, Sniehotta F, Schuz B. Predicting binge-drinking behaviour using an extended TPB: examining the impact of anticipated regret and descriptive norms. Alcohol Alcohol. 2007 Mar-Apr;42(2):84-91. doi: 10.1093/alcalc/agl115. Epub 2006 Dec 21. PMID 17185302
- [Background] Coolidge T, Skaret E, Heima M, Johnson EK, Hillstead MB, Farjo N, Asmyhr O, Weinstein P. Thinking about going to the dentist: a Contemplation Ladder to assess dentally-avoidant individuals' readiness to go to a dentist. BMC Oral Health. 2011 Jan 27;11:4. doi: 10.1186/1472-6831-11-4. PMID 21272356
- [Background] Epstude K, Roese NJ. The functional theory of counterfactual thinking. Pers Soc Psychol Rev. 2008 May;12(2):168-92. doi: 10.1177/1088868308316091. PMID 18453477
- [Background] Hogue A, Dauber S, Morgenstern J. Validation of a contemplation ladder in an adult substance use disorder sample. Psychol Addict Behav. 2010 Mar;24(1):137-44. doi: 10.1037/a0017895. PMID 20307121
- [Background] McGee R, Williams S, Kypri K. College students' readiness to reduce binge drinking: criterion validity of a brief measure. Drug Alcohol Depend. 2010 Jun 1;109(1-3):236-8. doi: 10.1016/j.drugalcdep.2009.12.009. Epub 2010 Jan 27. PMID 20106607
- [Background] Roese, N. J., Epstude, K. (2017). The functional theory of counterfactual thinking: New evidence, new challenges, new insights. Advances in Experimental Social Psychology, 56, 1-79.
- [Background] Smallman R, Roese NJ. Counterfactual Thinking Facilitates Behavioral Intentions. J Exp Soc Psychol. 2009 Jul;45(4):845-852. doi: 10.1016/j.jesp.2009.03.002. PMID 20161221
- [Background] Tal-Or, N., Boninger, D. S., & Gleicher, F. (2004). On becoming what we might have been: Counterfactual thinking and self-efficacy. Self and Identity, 3(1), 5-26.
- [Background] Wong, E. M. (2007). Narrating near-histories: The effects of counterfactual communication on motivation and performance. Management & Organizational History, 2(4), 351-370. https://doi.org/10.1177/1744935907086119

DOCUMENTS (4):
  • Study Protocol (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT05208593/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT05208593/SAP_001.pdf
  • Informed Consent Form: Consent for Baseline Session (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT05208593/ICF_002.pdf
  • Informed Consent Form: Consent for Follow-Up Sessions (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT05208593/ICF_003.pdf